CLINICAL TRIAL: NCT04638049
Title: Intestinal Microbiota in Prostate Cancer Patients as a Biomarker for Radiation-INduced Toxicity (IMPRINT): A Prospective Biomarker Study
Brief Title: Intestinal Microbiota in Prostate Cancer Patients as a Biomarker for Radiation-INduced Toxicity (IMPRINT)
Acronym: IMPRINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BC-07902
Record Dates: First submitted 2020-10-30; First posted 2020-11-20 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2020-10

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Prostatic Neoplasms
Keywords: Radiotherapy; Microbiome; Metabolome
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prostate (Bed) only RadioTherapy (PBRT) (Active Comparator): Primary, adjuvant or salvage RT of the prostate (bed) without RT of the pelvic nodal regions in the small pelvis, according to local hospital guidelines and protocols.
  Interventions: Other: Collection of human biofluids; Other: Patient reported outcome measures
- Whole Pelvis RadioTherapy (WPRT) (Active Comparator): Primary, adjuvant or salvage RT of the pelvic nodal regions in the small pelvis with possible additional RT of the prostate (bed), according to local hospital guidelines and protocols.
  Interventions: Other: Collection of human biofluids; Other: Patient reported outcome measures

INTERVENTIONS:
Other: Collection of human biofluids — Feces, blood and urine: (1) shortly before, (2) during and (3) shortly after RT treatment, as well as (4) one-month post-RT
Other: Patient reported outcome measures — EORTC QLQ-C30, PR25: (1) shortly before and (2) shortly after RT treatment, as well as (3) one-month post-RT

SUMMARY:
Radiotherapy (RT) of the abdomen and/or pelvis is known to cause acute and late gastrointestinal (GI) toxicities. While radiation dose and volume are known risk factors for developing such side effects, recent evidence suggests patterns of disturbance in the composition of the GI microbiota - so called "dysbiosis" - may also promote the host's susceptibility to GI toxicities through impaired intestinal barrier function and inflammation. The IMPRINT-study aims to expand the current knowledge on the role of intestinal bacteria and their metabolites involved in the pathophysiology of radiation-induced GI toxicities by longitudinally examining the microbiota composition (feces), the associated metabolome (blood, feces and urine) and bacterial extracellular vesicles (BEVs) (blood and feces).

DETAILED DESCRIPTION:
The IMPRINT-study is a prospective biomarker study assessing the impact of different treatment field sizes and associated radiation doses on the patient's microbiome and metabolome, whereby the link with radiation-induced GI toxicities will be emphasized. Blood, urine and fecal samples will be longitudinally collected at 4 different time points: (1) shortly before, (2) during and (3) shortly after RT treatment, as well as (4) one-month post-RT. To our knowledge, this is the first clinical research project relating the impact of multiple radiation parameters on fecal-, urine- and blood-based biomarkers to risk of GI toxicities in a homogeneously defined study population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven (initial) adenocarcinoma of the prostate
* Localized (confined to primary site) and/or regional (spread to regional pelvic lymph nodes) disease stage at diagnosis
* Age ≥ 18 years
* RT is an integral part of the treatment - primary, adjuvant or salvage
* WHO performance status 0-2
* Administration of androgen deprivation therapy (ADT) before RT
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Signed informed consent form (ICF) according to ICH/GCP and national/regional regulations

Exclusion Criteria:

* Other primary tumor (except for non-melanoma skin cancer) diagnosed < 5 years before enrollment
* Diagnosis of inflammatory bowel disease (e.g. Crohn's disease or ulcerative colitis)
* Administration of systemic therapy during RT other that ADT
* Subjected to antibiotic treatment or medically imposed dietary restrictions < 1 month prior to enrollment
* Body mass index (BMI) > 35
* Administration of pelvic RT < 1 year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Microbiome profiles as assessed by fecal samples | Up to 3.5 months after inclusion
  Characterization of dynamic changes in the intestinal microbiota composition using 16S rRNA sequencing technology
Metabolome profiles as assessed by fecal, blood and urine samples | Up to 3.5 months after inclusion
  Characterization of dynamic changes in the concentration of all small molecules (metabolites) in feces, blood and urine using ultra-high performance liquid chromatography coupled to high-resolution mass spectrometry (UHPLC-HRMS)

SECONDARY OUTCOMES:
Discovery of potential predictive biomarkers for the development of RT-induced GI toxicities | Up to 3.5 months after inclusion
  The identified microbiota and metabolite signatures will be investigated for association with incidence and severity of GI toxicities
Incidence of GI and Genitourinary (GU) toxicities | Up to 3.5 months after inclusion
  GI and GU toxicities as per Common Terminology for Adverse Events (CTCAE) v4.0
Patient reported QOL as per EORTC-QLQ C30 | Up to 3.5 months after inclusion
  Validated questionnaire assessing different health-related parameters (psychological, physical and social well-being) in cancer patients
Patient reported QOL as per EORTC-QLQ PR25 | Up to 3.5 months after inclusion
  Validated questionnaire assessing the health-related QOL of prostate cancer patients
Concentration of BEVs in fecal and blood samples | Up to 3.5 months after inclusion
  BEVs in fecal and blood samples will be separated and analyzed through the orthogonal implementation of ultrafiltration, size-exclusion chromatography (SEC) and density-gradient centrifugation, followed by biochemical characterization

CONTACTS AND LOCATIONS:
Overall Officials: Piet Ost, MD, PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium